CLINICAL TRIAL: NCT02389894
Title: Neuroprotection In Patients Undergoing Aortic Valve Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Annetine Gelijns, Chair, Department of Population Health Science & Policy, Edmond A. Guggenheim Professor of Health Policy Co-Director, InCHOIR, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GCO 08-1078-0009; 2U01HL088942-07 (NIH)
Record Dates: First submitted 2015-03-10; First posted 2015-03-17 (Estimated); Results first posted 2019-04-29 (Actual); Last update posted 2019-04-29 (Actual); Status verified 2019-04

CONDITIONS: Aortic Stenosis; Brain Infarction; Cerebrovascular Accident; Stroke
Keywords: Embolic Protection Device; Stroke; Brain Infarction; atheroma; Aortic Valve Replacement
MeSH Terms: conditions — Aortic Valve Stenosis; Brain Infarction; Stroke; Plaque, Atherosclerotic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Embol-X Embolic Protection Device (Active Comparator): The surgeon may use either the EMBOL-X® Access Device/Aortic Cannula or a standard cannula with the EMBOL-X® filter deployed through a separate introducer sheath.
  Interventions: Device: Embol-X Embolic Protection Device
- CardioGard Cannula (Active Comparator): The Cardiogard embolic protection device is a curved tip 24-French aortic perfusion cannula.
  Interventions: Device: CardioGard Cannula
- Standard Cannula (No Intervention): Patients in this arm will receive the standard of care surgical procedure using a cannula of the surgeon's choosing.

INTERVENTIONS:
Device: Embol-X Embolic Protection Device — per the manufacturer's instructions for use (IFU).
  Other Names: Edwards Embol-X embolic protection device
  Arms: Embol-X Embolic Protection Device
Device: CardioGard Cannula — CardioGard Cannula, per the manufacturer's instructions for use (IFU).
  Other Names: CardioGard Emboli Protection Cannula
  Arms: CardioGard Cannula

SUMMARY:
To evaluate the efficacy and safety of embolic protection devices to reduce ischemic brain injury in patients undergoing surgical aortic valve replacement (AVR).

DETAILED DESCRIPTION:
This is a multicenter randomized trial in which patients diagnosed with calcific aortic stenosis (AS) with planned AVR will be randomized to 1) the treatment arm of the Edwards Life Science filter and cannula or the filter as a stand alone with any cannula or 2) to the treatment arm of the CardioGard cannula versus 3) standard care in a 1:1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years
* Planned and scheduled surgical aortic valve replacement via a full or minimal-access sternotomy (using central aortic perfusion cannulae) for calcific aortic stenosis with a legally marketed valve
* No evidence of neurological impairment as defined by a NIHSS ≤1 and modified Rankin scale (mRS) ≤ 2 within 7 days prior to randomization
* Ability to provide informed consent and comply with the protocol

Exclusion Criteria:

* Contraindication to legally marketed embolic protection devices (e.g. aneurysm of the ascending aorta, aortic trauma, porcelain aorta, known sensitivity to heparin)
* History of clinical stroke within 3 months prior to randomization
* Cardiac catheterization within 3 days of the planned aortic valve replacement
* Cerebral and or aortic arch arteriography or interventions within 3 days of the planned aortic valve replacement
* Active endocarditis at time of randomization
* Anticipated inability to tolerate or contraindication for MRI (e.g., known intolerance of MRI, permanent pacemaker at baseline or expected implantation of a permanent pacemaker)
* Any other concomitant aortic procedure such as root replacement
* Concomitant surgical procedures other than CABG, mitral annuloplasty, left atrial appendage (LAA) excision or exclusion, atrial septal defect (ASD) closure or patent foramen ovale (PFO) closure
* Clinical signs of cardiogenic shock or treatment with IV inotropic therapy prior to randomization
* Concurrent participation in an interventional (drug or device) trial

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 383 (Actual)
Dates: Start 2015-03; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Annetine C Gelijns, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Richard Weisel, MD, Study Chair — Toronto General Hospital
Locations (18):
- United States (14):
  - University of Southern California, Los Angeles, California
  - Emory University, Atlanta, Georgia
  - University of Maryland, Baltimore, Maryland
  - NIH Heart Center at Suburban Hospital, Bethesda, Maryland
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Columbia University Medical Center, New York, New York
  - Montefiore Einstein Heart Center, The Bronx, New York
  - Mission Hospital, Asheville, North Carolina
  - Duke University, Durham, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Baylor Research Institute, Plano, Texas
  - University of Virginia, Charlottesville, Virginia
- Canada (4):
  - University of Alberta Hospital, Edmonton, Alberta
  - Toronto General Hospital, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - Institut Universitaire de Cardiologie de Quebec (Hopital Laval), Québec, Quebec

REFERENCES:
- [Derived] Messe SR, Overbey JR, Thourani VH, Moskowitz AJ, Gelijns AC, Groh MA, Mack MJ, Ailawadi G, Furie KL, Southerland AM, James ML, Moy CS, Gupta L, Voisine P, Perrault LP, Bowdish ME, Gillinov AM, O'Gara PT, Ouzounian M, Whitson BA, Mullen JC, Miller MA, Gammie JS, Pan S, Erus G, Browndyke JN; Cardiothoracic Surgical Trials Network (CTSN) Investigators. The impact of perioperative stroke and delirium on outcomes after surgical aortic valve replacement. J Thorac Cardiovasc Surg. 2024 Feb;167(2):624-633.e4. doi: 10.1016/j.jtcvs.2022.01.053. Epub 2022 Mar 18. PMID 35483981
- [Derived] Crestanello JA. "Not in my brain": The use of embolic protection devices to prevent brain embolization during cardiovascular procedures. J Thorac Cardiovasc Surg. 2018 Dec;156(6):e205-e206. doi: 10.1016/j.jtcvs.2018.05.114. Epub 2018 Jun 23. No abstract available. PMID 30007783
- [Derived] Mack MJ, Acker MA, Gelijns AC, Overbey JR, Parides MK, Browndyke JN, Groh MA, Moskowitz AJ, Jeffries NO, Ailawadi G, Thourani VH, Moquete EG, Iribarne A, Voisine P, Perrault LP, Bowdish ME, Bilello M, Davatzikos C, Mangusan RF, Winkle RA, Smith PK, Michler RE, Miller MA, O'Sullivan KL, Taddei-Peters WC, Rose EA, Weisel RD, Furie KL, Bagiella E, Moy CS, O'Gara PT, Messe SR; Cardiothoracic Surgical Trials Network (CTSN). Effect of Cerebral Embolic Protection Devices on CNS Infarction in Surgical Aortic Valve Replacement: A Randomized Clinical Trial. JAMA. 2017 Aug 8;318(6):536-547. doi: 10.1001/jama.2017.9479. PMID 28787505

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Embol-X Embolic Protection Device | CardioGard Cannula | Standard Cannula
Started | 133 | 118 | 132
Completed | 125 | 108 | 123
Not Completed | 8 | 10 | 9
Not completed — Death | 4 | 5 | 3
Not completed — Withdrawal by Subject | 2 | 4 | 5
Not completed — Lost to Follow-up | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Embol-X Embolic Protection Device | CardioGard Cannula | Standard Cannula | Total
Number analyzed (Participants) | 133 | 118 | 132 | 383
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.6 (6.6) | 74.6 (6.8) | 73.6 (6.7) | 73.9 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 49 | 46 | 147
  Male | 81 | 69 | 86 | 236
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 8 | 17
  Not Hispanic or Latino | 127 | 110 | 121 | 358
  Unknown or Not Reported | 2 | 3 | 3 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 2
  Asian | 0 | 0 | 5 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 7 | 6 | 19
  White | 126 | 108 | 118 | 352
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  Canada | 19 | 19 | 19 | 57
  United States | 114 | 99 | 113 | 326

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Freedom From Clinical or Radiographic Central Nervous System (CNS) Infarction
Description: freedom from CNS infarction, defined as brain, spinal cord, or retinal cell death attributable to ischemia based on neuropathological, neuroimaging, or clinical evidence of permanent injury based on symptoms persisting > 24 hours, with overt symptoms or no known symptoms. All patients will be assessed by 1.5 T (3.0 T is acceptable if 1.5 T not available) Diffusion-weighted imaging (DWI) at 7 (± 3) days post procedure for presence of brain lesions and to measure the number and volume of any present lesions.
Time Frame: up to 10 days post procedure
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Embol-X Embolic Protection Device | CardioGard Cannula | Standard Cannula
Number analyzed (Participants) | 133 | 118 | 132
percentage of participants | 74.4 [66.4 to 82.5] | 68.0 [59.1 to 76.8] | 67.6 [58.8 to 76.4]
Statistical Analysis 1: Comparison: Embol-X Embolic Protection Device vs Standard Cannula; A sample size of 165 patients in each group ensured that each comparison had a power of approximately 90% to detect a between-group difference of 17.5% from an assumed control rate of 50% in the incidence of postoperative CNS infarcts. A single interim analysis was prespecified and performed. Based on the recommendation of the DSMB, randomization but not follow-up was halted due to low conditional power of observing any between-group differences for the primary endpoint; Test type: Superiority; p = 0.22, Chi-squared; The primary end point analysis used an iterative hot-deck multiple imputation approach, assuming a nonignorable missing data mechanism; Risk Difference (RD) = 6.9, 95% CI 2-sided [-4.2 to 17.9] — The absolute difference in the percentage of patients with freedom from clinical or radiographic central nervous system (CNS) infarction was computed as Embol-x minus control
Statistical Analysis 2: Comparison: CardioGard Cannula vs Standard Cannula; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.84, Chi-squared — The primary end point analysis used an iterative hot-deck multiple imputation approach, assuming a nonignorable missing data mechanism; Risk Difference (RD) = 1.3, 95% CI 2-sided [-11.2 to 13.8] — The absolute difference in the percentage of patients with freedom from clinical or radiographic central nervous system (CNS) infarction was computed as Cardiogard minus control

2. Secondary Outcome: Number of Participants With a Composite Endpoint of Mortality, Clinical Stroke, and Acute Kidney Injury
Description: The number of patients who have had a clinical ischemic stroke, acute kidney injury (AKI), or death within 30 days of surgery.
Time Frame: up to 30 days
Population: Three patients withdrew prior to day 30 and are not included in the denominators
Measure: Count of Participants; unit: Participants
Arm/Group | Embol-X Embolic Protection Device | CardioGard Cannula | Standard Cannula
Number analyzed (Participants) | 132 | 117 | 131
Participants | 44 | 25 | 31
Statistical Analysis 1: Comparison: Embol-X Embolic Protection Device vs CardioGard Cannula; Test type: Superiority; p = 0.08, Chi-squared; Risk Difference (RD) = 9.7, 95% CI 2-sided [-1.2 to 20.5] — The absolute difference was computed as Embol-x minus control
Statistical Analysis 2: Comparison: CardioGard Cannula vs Standard Cannula; Test type: Superiority; p = 0.61, Chi-squared; Risk Difference (RD) = -2.8, 95% CI 2-sided [-13.5 to 7.9] — The absolute difference was computed as Cardiogard minus control

3. Secondary Outcome: Number of Patients With Clinically Apparent Stroke at 7 Days
Description: The number of patients who experience a clinically apparent stroke by 7 days post-op
Time Frame: at 7 days
Population: Two patients withdrew prior to day 7
Measure: Count of Participants; unit: Participants
Arm/Group | Embol-X Embolic Protection Device | CardioGard Cannula | Standard Cannula
Number analyzed (Participants) | 133 | 117 | 131
Participants | 11 | 6 | 8

4. Secondary Outcome: Presence of Radiographic Infarcts
Description: The proportion of patients with radiographic infarcts on day 7 (+/-3 days) MRI. Presences of radiographic infarcts were measured using diffusion-weighted 1.5 or 3T MRI scanners
Time Frame: up to 10 days
Population: Denominator includes all patients with day 7 MRI
Measure: Count of Participants; unit: Participants
Arm/Group | Embol-X Embolic Protection Device | CardioGard Cannula | Standard Cannula
Number analyzed (Participants) | 115 | 101 | 118
Participants | 83 | 66 | 76

5. Secondary Outcome: Total Infarct Volume
Description: Total infarct volume measured on day 7 dwMRI.
Time Frame: Day 7
Population: Analysis population includes all those with dwMRI at 7 days
Measure: Median (Inter-Quartile Range); unit: mm^3
Arm/Group | Embol-X Embolic Protection Device | CardioGard Cannula | Standard Cannula
Number analyzed (Participants) | 115 | 101 | 118
mm^3 | 74 [0 to 322] | 42 [0 to 151] | 35 [0 to 168]

6. Secondary Outcome: Decline in Overall Neurocognition
Description: Decline in neurocognitive function at 90 days as compared to baseline. Decline defined as the number of patients whose Z score (computed relative to the study population at baseline, adjusting for age, education and sex) at day 90 had decreased by 0.5 SD relative to the baseline score.
Time Frame: baseline and 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Embol-X Embolic Protection Device | CardioGard Cannula | Standard Cannula
Number analyzed (Participants) | 98 | 81 | 96
Participants | 28 | 24 | 31

7. Secondary Outcome: Decline in Neurocognitive Function in the Verbal Memory Domain at 90 Days
Description: Decline in neurocognitive function in the verbal memory domain at 90 days as compared to baseline. Decline defined as the number of patients whose Z score (computed relative to the study population at baseline, adjusting for age, education and sex) at day 90 had decreased by 0.5 SD relative to the baseline score.
Time Frame: baseline and 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Embol-X Embolic Protection Device | CardioGard Cannula | Standard Cannula
Number analyzed (Participants) | 117 | 94 | 111
Participants | 31 | 38 | 35

8. Secondary Outcome: Decline in Neurocognitive Function in the Visual Memory Domain at 90 Days
Description: Decline in neurocognitive function in the visual memory domain at 90 days as compared to baseline. Decline defined as the number of patients whose Z score (computed relative to the study population at baseline, adjusting for age, education and sex) at day 90 had decreased by 0.5 SD relative to the baseline score.
Time Frame: baseline and 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Embol-X Embolic Protection Device | CardioGard Cannula | Standard Cannula
Number analyzed (Participants) | 116 | 95 | 112
Participants | 36 | 25 | 32

9. Secondary Outcome: Decline in Neurocognitive Function in the Executive Function Domain at 90 Day
Description: Decline in neurocognitive function in the executive function domain at 90 days as compared to baseline. Decline defined as the number of patients whose Z score (computed relative to the study population at baseline, adjusting for age, education and sex) at day 90 had decreased by 0.5 SD relative to the baseline score.
Time Frame: baseline and 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Embol-X Embolic Protection Device | CardioGard Cannula | Standard Cannula
Number analyzed (Participants) | 103 | 83 | 99
Participants | 19 | 25 | 31

10. Secondary Outcome: Decline in Neurocognitive Function in the Visuospatial/Constructional Praxis Domain at 90 Days
Description: Decline in neurocognitive function in the visuospatial/constructional praxis domain at 90 days as compared to baseline. Decline defined as the number of patients whose Z score (computed relative to the study population at baseline, adjusting for age, education and sex) at day 90 had decreased by 0.5 SD relative to the baseline score.
Time Frame: baseline and 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Embol-X Embolic Protection Device | CardioGard Cannula | Standard Cannula
Number analyzed (Participants) | 117 | 98 | 113
Participants | 31 | 28 | 41

11. Secondary Outcome: Decline in Neurocognitive Function in the Auditory-Verbal Simple Attention Domain at 90 Days
Description: Decline in neurocognitive function in the Auditory-Verbal Simple attention domain at 90 days as compared to baseline. Decline defined as the number of patients whose Z score (computed relative to the study population at baseline, adjusting for age, education and sex) at day 90 had decreased by 0.5 SD relative to the baseline score.
Time Frame: baseline and 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Embol-X Embolic Protection Device | CardioGard Cannula | Standard Cannula
Number analyzed (Participants) | 117 | 96 | 112
Participants | 36 | 28 | 38

12. Secondary Outcome: Decline in Neurocognitive Function in the Visuomotor/Information Processing Speed Domain at 90 Days
Description: Decline in neurocognitive function in the Visuomotor/Information Processing Speed domain at 90 days as compared to baseline. Decline defined as the number of patients whose Z score (computed relative to the study population at baseline, adjusting for age, education and sex) at day 90 had decreased by 0.5 SD relative to the baseline score.
Time Frame: baseline and 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Embol-X Embolic Protection Device | CardioGard Cannula | Standard Cannula
Number analyzed (Participants) | 110 | 93 | 108
Participants | 43 | 30 | 33

13. Secondary Outcome: Modified Rankin Scale >2 at 90 Days
Description: The scale runs from 0-6, running from perfect health without symptoms to death. 0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Dead.
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Embol-X Embolic Protection Device | CardioGard Cannula | Standard Cannula
Number analyzed (Participants) | 127 | 110 | 123
Participants | 5 | 7 | 5

14. Secondary Outcome: Barthel Index <= 80
Description: An overall score has full range from 0 to 100, with higher scores indicating greater independence.
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Embol-X Embolic Protection Device | CardioGard Cannula | Standard Cannula
Number analyzed (Participants) | 123 | 105 | 120
Participants | 2 | 2 | 4

15. Secondary Outcome: Number of Participants With Confusion Assessment Method (CAM) Delirium Assessment at 7 Days
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Embol-X Embolic Protection Device | CardioGard Cannula | Standard Cannula
Number analyzed (Participants) | 123 | 112 | 122
Participants | 10 | 7 | 19

16. Secondary Outcome: Mortality by 90 Days
Description: Incidence of all-cause mortality
Time Frame: up to 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Embol-X Embolic Protection Device | CardioGard Cannula | Standard Cannula
Number analyzed (Participants) | 133 | 118 | 132
Participants | 4 | 5 | 3

17. Secondary Outcome: Length of Stay for Index Hospitalization
Time Frame: up to 90 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Embol-X Embolic Protection Device | CardioGard Cannula | Standard Cannula
Number analyzed (Participants) | 133 | 117 | 131
days | 10.4 (7.0) | 9.8 (6.7) | 10.3 (6.2)

18. Secondary Outcome: Hospital Readmissions
Description: Rate of hospital readmissions
Time Frame: up to 90 days
Measure: Number; unit: rate per 100-patient-months
Arm/Group | Embol-X Embolic Protection Device | CardioGard Cannula | Standard Cannula
Number analyzed (Participants) | 133 | 117 | 131
rate per 100-patient-months | 9.3 | 8.4 | 7.1

19. Secondary Outcome: Quality of Life - Physical Health Composite
Description: Quality of Life - Physical Health Composite Assessed by Short Form-12 (SF-12). Score ranking from 0 (worst health) to 100 (best health) calculated as the weighted sum of the questions. health scores then transformed into a t-score on the assumption that each question carries equal weight and were standardized to have mean of 50 and standard deviation of 10.
Time Frame: at 90 days
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Embol-X Embolic Protection Device | CardioGard Cannula | Standard Cannula
Number analyzed (Participants) | 122 | 102 | 119
T-Score | 43.0 (10.8) | 44.9 (8.3) | 44.2 (9.0)

20. Secondary Outcome: Quality of Life - Mental Health Composite
Description: Quality of life - Mental health composite Assessed by Short Form-12 (SF-12). Score ranking from 0 (worst health) to 100 (best health) calculated as the weighted sum of the questions. health scores then transformed into a t-score on the assumption that each question carries equal weight and were standardized to have mean of 50 and standard deviation of 10.
Time Frame: at 90 days
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Embol-X Embolic Protection Device | CardioGard Cannula | Standard Cannula
Number analyzed (Participants) | 122 | 102 | 119
T-Score | 55.2 (10.2) | 55.4 (8.2) | 54.8 (8.0)

21. Secondary Outcome: Number of Participants With Emboli Captured
Description: Assessed by the presence of any debris captured in filter of embolic protection device
Time Frame: day 1
Population: Emboli are not captured by the standard cannula and therefore no data are available for this group in this outcome measure
Measure: Count of Participants; unit: Participants
Arm/Group | Embol-X Embolic Protection Device | CardioGard Cannula | Standard Cannula
Number analyzed (Participants) | 116 | 106 | 0
Participants | 115 | 79 | 0

ADVERSE EVENTS:
Time Frame: 90 Days
Arm/Group | Embol-X Embolic Protection Device | CardioGard Cannula | Standard Cannula
All-Cause Mortality (participants affected / at risk) | 4/133 | 5/118 | 3/132
Serious Adverse Events (participants affected / at risk) | 72/133 | 53/118 | 54/132
Other Adverse Events (participants affected / at risk) | 45/133 | 47/118 | 43/132
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Embol-X Embolic Protection Device (N=133) | CardioGard Cannula (N=118) | Standard Cannula (N=132)
Acute Kidney Injury - Stage 1 (Renal and urinary disorders) | 3 (3) | 1 (1) | 0 (0)
Acute Kidney Injury - Stage 2 (Renal and urinary disorders) | 4 (4) | 0 (0) | 2 (2)
Acute Kidney Injury - Stage 3 (Renal and urinary disorders) | 7 (7) | 2 (2) | 2 (2)
Bleeding - Transfusion > 5 units RBC <24 hours following surgery (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Bleeding - Re-operation for hemorrhage or tamponade (Blood and lymphatic system disorders) | 5 (5) | 7 (7) | 5 (5)
Cardiac Arrhythmias - Cardiac arrest (Cardiac disorders) | 5 (6) | 0 (0) | 2 (2)
Cardiac Arrhythmias - Sustained ventricular arrhythmia requiring defibrillation or cardioversion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac Arrhythmias - Sustained supraventricular arrhythmia requiring drug treatment or cardioversio (Cardiac disorders) | 42 (43) | 22 (25) | 25 (25)
Cardiac Arrhythmias - Cardiac conduction abnormalities or sustained bradycardia requiring permanent (Cardiac disorders) | 7 (7) | 6 (6) | 3 (3)
Pericardial Fluid Collection (Cardiac disorders) | 4 (4) | 1 (1) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 12 (14) | 10 (13) | 9 (11)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 3 (3)
Hepatic Dysfunction (Liver injury and Impaired Liver function) (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Major Infection - Localized Infection (Infections and infestations) | 13 (14) | 7 (7) | 10 (11)
Major Infection - Endocarditis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Major Infection - Sepsis (Infections and infestations) | 1 (1) | 2 (2) | 4 (4)
Myocardial Infarction - Non-Procedure Related (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial Infarction - Peri-CABG (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Neurological Dysfunction- Transient Ischemic Attack - TIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Neurological Dysfunction- Ischemic Stroke (Nervous system disorders) | 3 (4) | 3 (3) | 4 (4)
Neurological Dysfunction- Toxic Metabolic Encephalopathy (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1)
Neurological Dysfunction- Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3)
Neurological Dysfunction- Other Neurological Dysfunction* (Nervous system disorders) | 1 (1) | 0 (0) | 3 (3)
Renal Events (Renal Failure) (Renal and urinary disorders) | 1 (1) | 0 (0) | 2 (2)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 3 (3) | 10 (11)
Heart Failure (Cardiac disorders) | 2 (2) | 4 (4) | 8 (9)
Venous Thromboembolism Event - Deep Vein Thrombosis (Vascular disorders) | 2 (3) | 0 (0) | 2 (2)
Venous Thromboembolism Event - Pulmonary Embolism (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Venous Thromboembolism Event - Other* (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Wound Dehiscence (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0)
Adrenal Insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Aortic Valve Re-operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Chest Pain (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Dysphagia with PEG tube placement (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Fever (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fluid Overload (General disorders) | 1 (1) | 0 (0) | 0 (0)
Foot Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
GI Bleed (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2)
Hemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Hypertension (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Intra abdominal bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Lung mass (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Orthostatic Hypertension (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumoperitoneum (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Post-pericardiotomy Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Repair of Aorta (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Severe TR requiring TV replacement (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Small bowel obstruction/ileus (Gastrointestinal disorders) | 2 (2) | 0 (0) | 4 (4)
Syncope (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Weakness (General disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Embol-X Embolic Protection Device (N=133) | CardioGard Cannula (N=118) | Standard Cannula (N=132)
Acute Kidney Injury - Stage 1 (Renal and urinary disorders) | 21 (22) | 13 (13) | 21 (21)
Cardiac Arrhythmias - Sustained supraventricular arrhythmia requiring drug treatment or cardioversio (Cardiac disorders) | 23 (24) | 34 (34) | 24 (24)
Major Infection - Localized Infection (Infections and infestations) | 8 (9) | 6 (7) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No